CLINICAL TRIAL: NCT04094350
Title: Effect of Community Active Case Finding Strategies for Detection of Tuberculosis in Cambodia: Study Protocol for a Pragmatic Cluster Randomized Controlled Trial
Brief Title: Effect of Community Active Case Finding Strategies for Detection of Tuberculosis in Cambodia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: KHANA Center for Population Health Research (Other)
Responsible Party: Principal Investigator, Siyan Yi, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NIHA-2018-005
Record Dates: First submitted 2019-08-02; First posted 2019-09-18 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Community health services; Cambodia; Contact tracing; Mass screening; Referral and consultation; Peer group
MeSH Terms: conditions — Tuberculosis | interventions — A1CF protein, human

STUDY DESIGN:
Intervention Model Description: A 12-moth pragmatic cluster randomized controlled trial will be conducted to evaluate different TB case-finding strategies. Eights operational districts consisting a total of 70 health centers will be randomized into one of the four groups (2 operational district per group): 1) Active case finding (ACF) with the seed-and-recruit model by KHANA, 2) ACF targeting household and neighborhood contacts by the National Center for Tuberculosis and Leprosy Control (CENAT), 3) ACF targeting the older population using mobile screening units by Cambodia Anti-Tuberculosis Association (CATA) and 4) Passive case finding (PCF).
Who Masked: Outcomes Assessor
Masking Description: Project coordinators and residents in the selected operational districts will not be masked to the intervention. However, all case finding activities will be done without reference to the intervention group. The data analysts will be masked to intervention allocation and will only analyse de-identified data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ACF with a seed-and-recruit model (Experimental): Active case finding with a seed-and-recruit model to be implemented by KHANA. Target group: key populations for TB (people living with HIV, TB contacts, people with diabetes, people who use/inject drugs) and presumptive TB cases
  Interventions: Other: ACF targeting household and neighborhood contacts; Other: ACF targeting the older population using mobile screening units; Other: Passive case finding
- ACF targeting household and neighborhood contacts (Experimental): Active case finding targeting household and neighborhood contacts to be implemented by CENAT. Target group: household contacts, immediate neighbors of people diagnosed with TB in the last 2 years, and other presumptive TB cases
  Interventions: Other: ACF with a seed-and-recruit model
- ACF targeting the older population (Experimental): Active case finding targeting the older population (people aged 55 and older) using mobile screening units to be implemented by CATA. Target group: elderly above age of 55 and other presumptive TB cases
  Interventions: Other: ACF with a seed-and-recruit model
- Passive case finding (No Intervention): Passive case finding strategy is a default setup in the national health system. PCF relies on the self-presentation of presumptive TB cases to the health centers to be diagnosed with TB.

INTERVENTIONS:
Other: ACF with a seed-and-recruit model — The intervention will take place for 12 months. In the intervention clusters, potential seeds - TB survivors, people living with HIV, and household contacts of people with TB - will be approached by the research team. Seeds will be trained and act as recruiters in the community to refer presumptive TB cases to the attached health centers. The research team will work with staff at the health centers to facilitate screening and enrollment of recruits who are diagnosed with TB to care. New people with TB who have the potential to be a recruiter will be invited and trained to recruit their peers in the community who may have TB for TB screening. Seeds will be trained to identify people who may have TB and equipped with health promotion skills to impart knowledge and practices about TB. We will follow-up all people with TB referred by seeds for six months from the treatment initiation.
  Arms: ACF targeting household and neighborhood contacts; ACF targeting the older population
Other: ACF targeting household and neighborhood contacts — In this arm, community health volunteers will recruit household contacts of people with TB and TB survivors diagnosed during the preceding two years. Immediate neighbors (10 nearest households) of the index cases (people with TB) who are symptomatic will also be invited by the community health volunteers to the screening session. Next nearest households within the same village will be approached if the number of presumptive TB cases in the 10 nearest households is low. The one-off screening session will be held at the nearest health center on specific days. Presumptive TB cases will be screened for symptoms on-site, and chest x-ray (CXR) will be taken. Sputum samples from presumptive TB cases with abnormal (CXR) will be collected for GeneXpert testing. Test results will be communicated to the newly diagnosed people with TB, and they will be referred to the health centers for treatment and follow-up.
  Arms: ACF with a seed-and-recruit model
Other: ACF targeting the older population using mobile screening units — The outreach team will conduct training and sensitization of the target population of the activities. The schedule of a one-off screening session will be made known to the communities in the districts before the screening day. Each person who visits the screening session will be screened. Demographic information and presence of TB symptoms will be collected at registration by a trained staff. A chest x-ray will then be performed on-site for all persons exhibiting TB symptoms and all elderly aged 55 and above regardless of symptoms. When CXR findings are abnormal, sputum samples will be collected for GeneXpert testing on-site as well. Test results will be communicated to the participants on the spot or via phone calls, and people with TB will be referred for treatment and follow-up at the health center where screening is conducted or a center of their choice. Should the health center of their choice do not fall within the selected sites, follow-up will be conducted via phone calls.
  Arms: ACF with a seed-and-recruit model
Other: Passive case finding — Passive case finding (PCF) strategy is a default setup in the national health system. PCF relies on the self-presentation of presumptive TB cases to the health centers to be diagnosed with TB.
  Arms: ACF with a seed-and-recruit model

SUMMARY:
Tuberculosis (TB) is a highly stigmatized disease, and approximately one-third of the Cambodian population living with TB are undetected. Therefore, it is vital to find these missing cases and promptly link them to care to reduce disease progression and interrupt further transmission. The integration of community-based, peer-driven intervention in TB active case finding (ACF) is relatively novel. In partnership with KHANA, the National Center for Tuberculosis and Leprosy Control (CENAT), and the Cambodia Anti-Tuberculosis Association (CATA), we will conduct a pragmatic cluster randomized controlled trial comparing 1) the ACF with the seed-and-recruit model; 2) ACF targeting household and neighborhood contacts; 3) ACF targeting the older population using mobile screening units; and 4) passive case finding (PCF) approach. The primary outcome will be the case notification rate in the intervention and control districts during the study period. We will also determine additionality, comparing the yield in each arm with its respective historical baseline and the cumulative yield over the implementation period. The secondary outcomes include the number needed to screen to detect one TB case, cost-effectiveness (direct and indirect costs per TB case notified), and the treatment outcome of all people with TB in this study. The project will be carried out over two years in eight operational districts (province name in parenthesis) - Koh Soutin (Kampong Cham), Stong (Kampong Thom), Kanchreach (Prey Veng), Choeung Prey (Kampong Cham), Dambae (Thbong Khmum), Boribo (Kampong Chhnang), Ponhea Leu (Kandal), and Phnom Srouch (Kampong Speu) - in Cambodia. The selection was also based on the number of health centers to increase comparability and generalizability of study findings. This study will randomize currently underserved operational districts (without active intervention at least in the past six months from the implementation date) to receive the interventions (ACF) and PCF as the control. The results from this proposal will enable a nationwide scale-up of an effective intervention that is contextualized and complies with the principles set by the national TB program to find undiagnosed cases and control TB in Cambodia. Also, this project will complement existing ACF programs in Cambodia by expanding ACF to other operational districts that are currently not served by the Global Fund, its implementing partners, and other organizations. Findings from this trial could also potentially inform active case finding strategies in other countries with a high TB burden.

DETAILED DESCRIPTION:
Tuberculosis (TB) is a leading infectious cause of morbidity and mortality worldwide, accounting for 10 million new cases and 1.6 million deaths in 2017. The disease burden is disproportionately concentrated in low- and middle-income countries with over 95% of TB deaths contributed by these regions. In 2016, the number of new TB cases was estimated at 10 million, and nearly 40% remained undiagnosed. Limited access to health care, high treatment cost, and social stigma of TB contributed to delayed detection and poor treatment uptake. Other risk factors such as poor living conditions and overcrowding further perpetuated the transmission of TB, which, in turn, leads to social and economic insecurity. Cambodia is one of the countries with the world's highest burden of TB, with an estimated incidence of active TB of 326 (95% CI: 224-447) per 100,000 population in 2017. Through the years, TB control programs in Cambodia has achieved significant milestones made possible by committed partners and focused efforts at the grassroots, national, and international level. In 2016, the TB incidence was approximately half of that in the year 2000, and a similar decline was observed in the TB mortality rate. Furthermore, the country has made notable progress in the fight against TB by achieving a treatment success rate of 94%, one of the highest among the 30 high TB burden countries.

However, the successes are impeded by a significant proportion of undiagnosed cases. Globally, it is estimated that 36% of the TB cases were undiagnosed in 2017, and a similar proportion is observed in Cambodia. Traditionally, TB cases are captured and passively notified when people with TB present themselves to a health facility. In recent years, a more proactive strategy to increase TB case notification, namely active case finding (ACF) has gained traction and is reported to be effective. Alongside passive case finding (PCF), the ACF strategy has been adopted by countries affected by the epidemic, including Cambodia, to reach people with TB effectively. Nevertheless, despite increased efforts to improve case detection, TB case finding remains a great challenge due to limited resources, geographical barriers, and social stigma. The current approaches rely solely on skilled healthcare workers and community health volunteers to find TB cases. Its utility and sustainability, in the long run, have yet to be substantially demonstrated.

Empirically, a snowball approach (seed-and-recruit mechanism) has been widely accepted to reach concealed populations such as populations who are at-risk for HIV in many countries, including Cambodia, due to its practical feasibility. A community-based peer-led strategy as such has been an inherent component in HIV responses worldwide, and successes have been reported. However, little is known about the feasibility and effectiveness of ACF with the snowball model in improving TB case notification. However, given the comparable hard-to-reach nature of HIV and TB populations, it is a concept worth exploring. In partnership with KHANA, the National Center for Tuberculosis and Leprosy Control (CENAT), and the Cambodia Anti-Tuberculosis Association (CATA), this project seeks to examine the effectiveness of different ACF strategies in increasing TB case notification in the community and its impact on treatment outcome. This project is congruent with the global plan to end TB. and the Global Fund's strategy 2017-2022 by informing sustainable and evidence-based solutions for TB control in Cambodia.

We will conduct a cluster randomized controlled trial with four arms comparing ACF with the seed-and-recruit model, other ACF approaches, and PCF approach in eight operational districts in Cambodia. The project will be carried out over two years. ACF with the seed-and-recruit model by KHANA, ACF targeting household and neighborhood contacts by CENAT, ACF targeting the older population using mobile screening units by CATA will be implemented in the intervention arms and PCF will be implemented in the control arm. These case finding strategies have been piloted in Cambodia, and they are endorsed by the national TB program in Cambodia. This study will randomize currently underserved operational districts (without active intervention, at least in the past six months from the implementation date). The interventions will be carried out as per the protocol devised by the partner organizations, respectively.

This study aims to 1) evaluate the effectiveness of an ACF strategy using a seed-and-recruit model for increasing TB case notification (case notification rate, additionality, comparing the yield in each arm with its respective historical baseline and the cumulative yield over the implementation period) in Cambodia, 2) establish the effect of ACF strategies on TB treatment outcomes, 3) evaluate number needed to screen to detect one TB case and the cost-effectiveness (costs per TB case notified) of different ACF strategies.

ELIGIBILITY:
Inclusion Criteria:

Presumptive TB cases will be referred to the health centers for TB screening and diagnosis in the intervention arms and self-presented to the health centers in the control arm. We will include the aggregated number of cases diagnosed and notified from all arms regardless of age. In this project, an individual is defined as a presumptive TB case if he/she exhibits any of the following symptoms19:

1. Pulmonary TB (PTB): A cough more than two weeks and at least one general symptom
2. Extra-pulmonary TB (EPTB): Presence of symptoms, depending on the location of TB, (e.g., cervical lymph node, swollen backbone, swollen articulation, etc.) and at least one general symptom
3. General symptoms: Fever, night sweat for more than two weeks or unintentional weight loss (>5% reduction in usual body weight over the last 6 to 12 months)20

People newly diagnosed with TB age 18 and above* from the selected health centers. We will only include all people with TB aged 18 years or over with TB (all-forms) for the baseline and follow-up survey.

Exclusion Criteria:

* We will exclude those who refused to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2004 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Number of TB cases notified per 10000 population | During the intervention period (1 year)
  Number of TB cases notified per 10000 population by each operational district included in this study per year
Additional number of TB cases | During the intervention period (1 year)
  Additional number of TB cases reported compared to historical baseline (same period in the preceding 1 year)
Number of TB cases diagnosed per 1000 population screened | During the intervention period (1 year)
  Number of TB cases diagnosed per 1000 population screened during one year of the intervention period

SECONDARY OUTCOMES:
Number of people with TB who have completed TB treatment and successfully treated | Six months after TB treatment initiated
  Number of people with TB who have completed TB treatment and successfully treated 6 months after treatment initiation
Number of people needed to screen to detect one case | During the intervention period (1 year)
  Number needed to screen to detect one case = total number of presumptive TB cases screened / number of TB cases identified
Cost-effectiveness | During the intervention period (1 year)
  Cost per TB case diagnosed/notified and incremental cost-effectiveness ratio per disability-adjusted life year (DALY) averted

CONTACTS AND LOCATIONS:
Overall Officials: Siyan Yi, PhD, Principal Investigator — National University of Singapore; Alvin Teo, MPH, Principal Investigator — National University of Singapore
Locations (3):
- Cambodia (3):
  - KHANA Center for Population Health Research, Phnom Penh
  - Cambodia Anti-Tuberculosis Association, Phnom Penh
  - National Center for Tuberculosis and Leprosy Control, Phnom Penh

IPD SHARING:
Plan to Share IPD: No
IPD will be made available upon request due to ethics restriction.

REFERENCES:
- [Background] Kranzer K, Afnan-Holmes H, Tomlin K, Golub JE, Shapiro AE, Schaap A, Corbett EL, Lonnroth K, Glynn JR. The benefits to communities and individuals of screening for active tuberculosis disease: a systematic review. Int J Tuberc Lung Dis. 2013 Apr;17(4):432-46. doi: 10.5588/ijtld.12.0743. PMID 23485377
- [Background] Pascom AR, Szwarcwald CL, Barbosa Junior A. Sampling studies to estimate the HIV prevalence rate in female commercial sex workers. Braz J Infect Dis. 2010 Jul-Aug;14(4):385-97. PMID 20963326
- [Background] Simoni JM, Nelson KM, Franks JC, Yard SS, Lehavot K. Are peer interventions for HIV efficacious? A systematic review. AIDS Behav. 2011 Nov;15(8):1589-95. doi: 10.1007/s10461-011-9963-5. PMID 21598034
- [Background] Marton KI, Sox HC Jr, Krupp JR. Involuntary weight loss: diagnostic and prognostic significance. Ann Intern Med. 1981 Nov;95(5):568-74. doi: 10.7326/0003-4819-95-5-568. PMID 7294545
- [Result] GBD Tuberculosis Collaborators. The global burden of tuberculosis: results from the Global Burden of Disease Study 2015. Lancet Infect Dis. 2018 Mar;18(3):261-284. doi: 10.1016/S1473-3099(17)30703-X. Epub 2017 Dec 7. PMID 29223583
- [Result] Mhimbira FA, Cuevas LE, Dacombe R, Mkopi A, Sinclair D. Interventions to increase tuberculosis case detection at primary healthcare or community-level services. Cochrane Database Syst Rev. 2017 Nov 28;11(11):CD011432. doi: 10.1002/14651858.CD011432.pub2. PMID 29182800
- [Result] Eang MT, Satha P, Yadav RP, Morishita F, Nishikiori N, van-Maaren P, Weezenbeek CL. Early detection of tuberculosis through community-based active case finding in Cambodia. BMC Public Health. 2012 Jun 21;12:469. doi: 10.1186/1471-2458-12-469. PMID 22720878
- [Result] Morishita F, Eang MT, Nishikiori N, Yadav RP. Increased Case Notification through Active Case Finding of Tuberculosis among Household and Neighbourhood Contacts in Cambodia. PLoS One. 2016 Mar 1;11(3):e0150405. doi: 10.1371/journal.pone.0150405. eCollection 2016. PMID 26930415
- [Result] Murray EJ, Bond VA, Marais BJ, Godfrey-Faussett P, Ayles HM, Beyers N. High levels of vulnerability and anticipated stigma reduce the impetus for tuberculosis diagnosis in Cape Town, South Africa. Health Policy Plan. 2013 Jul;28(4):410-8. doi: 10.1093/heapol/czs072. Epub 2012 Sep 2. PMID 22945548
- [Result] Yaesoubi R, Cohen T. Identifying dynamic tuberculosis case-finding policies for HIV/TB coepidemics. Proc Natl Acad Sci U S A. 2013 Jun 4;110(23):9457-62. doi: 10.1073/pnas.1218770110. Epub 2013 May 20. PMID 23690585
- [Result] Koura KG, Trebucq A, Schwoebel V. Do active case-finding projects increase the number of tuberculosis cases notified at national level? Int J Tuberc Lung Dis. 2017 Jan 1;21(1):73-78. doi: 10.5588/ijtld.16.0653. PMID 28157468
- [Result] Yi S, Ngin C, Tuot S, Chhoun P, Chhim S, Pal K, Mun P, Mburu G. HIV prevalence, risky behaviors, and discrimination experiences among transgender women in Cambodia: descriptive findings from a national integrated biological and behavioral survey. BMC Int Health Hum Rights. 2017 May 23;17(1):14. doi: 10.1186/s12914-017-0122-6. PMID 28535758
- [Derived] Teo AKJ, Prem K, Evdokimov K, Ork C, Eng S, Tuot S, Chry M, Mao TE, Hsu LY, Yi S. Effect of community active case-finding strategies for detection of tuberculosis in Cambodia: study protocol for a pragmatic cluster randomized controlled trial. Trials. 2020 Feb 24;21(1):220. doi: 10.1186/s13063-020-4138-1. PMID 32093778